CLINICAL TRIAL: NCT05949216
Title: The Impact of Musical Engagement on Medical Resident Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Conor Donnelly (Other)
Responsible Party: Sponsor-Investigator, Conor Donnelly, Resident, Department of Family Medicine, McMaster University, McMaster University
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRM_Study
Record Dates: First submitted 2023-06-28; First posted 2023-07-17 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Burnout; Student Burnout; Physical Disability; Resident Doctor; Music Therapy; Music; Stress; Wellness, Psychological
MeSH Terms: conditions — Burnout, Psychological; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Musical engagement sessions (Experimental): The single group of this study will participate in four musical engagement sessions as described in the intervention section.
  Interventions: Behavioral: Musical engagement sessions

INTERVENTIONS:
Behavioral: Musical engagement sessions — Musical engagement sessions will be 2 hours long and involve improvisation and sight-reading of sheet music. Participants will supply their own instrument of choice to play. There will be four sessions total.

SUMMARY:
It is common knowledge that music has a positive impact on human well-being. It is also well-known that medical residents are frequently stressed and burnt out. With these two thoughts in mind, the investigators want to explore how participating in a musical engagement program may positively impact medical resident well-being. The investigators hope to do this by hosting four informal musical engagement sessions with medical residents, which will involve playing instruments, improvising, and reading sheet music. To study the impact that this program has on participants, investigators will ask participants to complete a survey. The investigators hope to find that participants are positively impacted by participation in the study, in terms of factors like stress reduction and minimized burnout symptoms. Hopefully, the study results may inform residency program curriculum designers in the future may incorporate music into wellness programming.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be residents in the Family Medicine program at McMaster University, in any year of study
2. Participants may be on any rotation in their program schedule and located at any site
3. Participants may be of any gender identity, age, ethnicity, and sexual orientation
4. Must identify as a "musician", whether casual, professional, or somewhere in between - however, they require enough musical training so that they may comfortably participate in the planned sight reading and improvisation within the study
5. Participants must be able to supply their own physical instrument for sessions
6. Must be aged 18 or over
7. Must be English-speaking

Exclusion Criteria:

1. Potential participant may not be a resident of any other residency program, or be from a university other than McMaster
2. If a participant is unable to participate in two or more musical sessions, they will not be included in this study
3. If a participant is unable to complete the qualitative and quantitative survey forms in their entirety, they will not be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Improvement of burnout symptoms | Eight weeks
  Participants will respond to three questionnaires - before, during, and after the study has completed. Questions will pertain to burnout symptoms and each will use a 5-point Likert scale. Options will be "strongly disagree", "disagree", "neutral", "agree", and "strongly disagree". Examples of questions include "I feel burnt out" and "I have difficulty concentrating at work". Questions will be identical between each questionnaire. By comparing answers between surveys we will be able to determine how burnout symptoms may have changed during the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No